CLINICAL TRIAL: NCT02824757
Title: Explore the Effects of Glucocorticoids on Glucose Metabolism by Continuous Glucose Monitoring in Patients With Interstitial Lung Disease
Brief Title: The Effects of Glucocorticoids on Glucose Metabolism in Patients With Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhao-ZS965
Record Dates: First submitted 2016-05-15; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Interstitial Lung Disease
Keywords: interstitial lung disease; glucocorticcoid; glucose; continuous glucose monitor
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- known diabetes: Participants have been diagnosed diabetes.
- known prediabetes: Participants have been diagnosed impaired glucose tolerance or impaired fasting glucose before.
- normal glucose tolerance: Participants have done the oral glucose tolerance test and been confirmed the normal glucose tolerance.
- unclear glucose tolerance condition: Participants who have not done oral glucose tolerance test or been diagnosed diabetes before.

SUMMARY:
This study is aimed at exploring the effects of glucocorticoids on glucose metabolism in patients with interstitial lung disease. Patients with interstitial lung disease who is on the medication of 15mg prednisolone and 7.5mg prednisolone conduct the continuous glucose monitoring (CGM). The data attained from the CGM are used to define the glycemic characteristics in patients using glucocorticoids and the difference of glucose features due to different doses.

DETAILED DESCRIPTION:
Patients diagnosed of interstitial lung disease and treating with glucocorticoids could be enrolled in this clinical trial. Those who is in an acute inflammatory phase and diagnosed with hemorrhagic disease should are excluded, so are those unwilling to carry the continuous glucose monitoring (CGM) device. When the dose of prednisolone is applied 15mg per day steadily and is going to be decreased, the CGM is conducted. At the same time, blood tests evaluating the glucose metabolism are measured, including HbA1c, GA, fasting insulin and fasting glucose. After taking 7.5mg prednisolone per day for 3 months, participants do the CGM and blood tests again to evaluate the glucose metabolism during this period. The CGM data could be used for the glucose evaluation, which can manifest the glucose characteristics in the circumstances of glucocorticoid use. By comparing the CGM data and the blood tests, the investigators hope to find the different features of the glucose metabolism due to different doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with interstitial lung disease

Exclusion Criteria:

* Patients who are in an acute inflammatory phase
* Patients who are diagnosed hemorrhagic disease
* Patients who are unwilling to carry the continuous glucose monitoring device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interstitial lung diseases(ILD), also known as diffuse parenchymal lung diseases, are a group of lung diseases with similar clinical, radiological and pathological manifestation. The causes include connective tissue disease-associated interstitial lung diseases, idiopathic interstitial pneumonias, granulomatous lung disorders etc. Most patients with ILD are recommended to take the glucocorticoid treatment. The adverse effects of glucocorticoids include the glucose metabolism disorder, weight gain, high blood pressure and osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The interstitial glucose values measured by CGMS (continuous glucose measure service) | 3 months
  A group of interstitial glucose values will be attained by the CGMS, the number of which count up to more than 1000. These data will undergo statistical process. CGM will be conducted twice when the participants take 15mg prednisolone stably and take 7.5mg prednisolone for 3 months. The difference between the two group of data will be evaluated and discussed.

SECONDARY OUTCOMES:
fasting insulin | 3 months
  The fasting insulin can evaluate the function of pancreatic beta cell to some extent. The fasting insulin will be evaluated twice when the participants take 15mg prednisolone stably and when the participants take 7.5mg prednisolone for 3 months.
fasting glucose | 3 months
  The fasting glucose could evaluate the glucose metabolism to some extent. The fasting glucose will be evaluated twice when the participants take 15mg prednisolone stably and when the participants take 7.5mg prednisolone for 3 months.
fasting C peptide | 3 months
  The fasting C peptide could evaluate the function of pancreatic beta cell to some extent. The fasting C peptide will be evaluated twice when the participants take 15mg prednisolone stably and when the participants take 7.5mg prednisolone for 3 months.
HbA1c | 3 months
  HbA1c could reflect the average blood glucose for 3 months. The HbA1c will be evaluated twice when the participants take 15mg prednisolone stably and when the participants take 7.5mg prednisolone for 3 months.
Glycated albumin | 3 months
  The glycated albumin could evaluate the average blood glucose in the previous 2 weeks to 1 month. The glycated albumin will be evaluated twice when the participants take 15mg prednisolone stably and when the participants take 7.5mg prednisolone for 3 months.

OTHER OUTCOMES:
Weight | 3 months
  The weight of each participant will be recorded to evaluate the weight change during the study.
waistline | 3 months
  The waistline of each participant will be recorded to evaluate the weight change during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Weigang Zhao, MD, Principal Investigator — Endocrinology department, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes